CLINICAL TRIAL: NCT06910020
Title: Effect of the Active Cycle of Breathing Technique on Coronary Artery Bypass Graft Patients' Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Shaimaa Nagi Abdelkader Yousef, Demonstrator of Critical Care and Emergency Nursing, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 320; 320 (Registry Identifier: Ethical Committee, Faculty of Nursing, Mansoura University)
Record Dates: First submitted 2025-03-18; First posted 2025-04-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Bypass; Coronary Arterial Disease (CAD)
Keywords: CABG; ACBT; Postoperative Pulmonary Complications; Chest tube duration; Hemodynamic parameters; Chest expansion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Cycle of Breathing Technique (Experimental): Patients who will perform ACBT exercises in addition to the routine ICU care.
  Interventions: Other: Active Cycle of Breathing Technique
- Control Group (No Intervention): Patients who will receive routine ICU care (chest physiotherapy and incentive spirometer) without ACBT.

INTERVENTIONS:
Other: Active Cycle of Breathing Technique — * Patients will assume the sitting position and relax their shoulders, then perform the following:
    1. Breathing control (abdominal breathing)
    2. Chest expansion (thoracic breathing)
    3. Huff cough (forced expiratory technique)
  * After completing the above actions, patients will be asked to cough up the residual deep sputum to promote pulmonary expansion.
  * The ACBT intervention will be performed for three days, each day two sessions, each session three courses, with 10 minutes of rest between them as needed.
  Arms: Active Cycle of Breathing Technique

SUMMARY:
Following CABG surgery, patients are at risk for several complications. One of the most common complications is postoperative pulmonary complications, which include atelectasis and dyspnea. These complications cause prolonged ICU length of stay and increased health care costs. Several studies recommended the active cycle of breathing technique as a method that increases secretion removal and improves lung functions, thus reducing the incidence of postoperative pulmonary complications. Our study aims to investigate the effect of the active cycle of breathing technique on coronary artery bypass graft patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who will undergo CABG

Exclusion Criteria:

* Mechanically ventilated patients on the first postoperative day.
* Patients with preoperative lung collapse or pleural effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Atelectasis | The first three postoperative days
  Atelectasis will be assessed using chest X-rays.
Dyspnea | The first three postoperative days
  Dyspnea level will be assessed using the modified Borg scale.
Functional capacity | The first three postoperative days
  Functional capacity will be assessed using the six-minute walk test
Hemodynamic parameters | The first three postoperative days
  Hemodynamic parameters will include respiratory rate expressed as the number of cycles per minute, which will be assessed using the cardiac monitor
Chest expansion | The first three postoperative days
  Chest expansion will be measured at three points (axillary, xiphoid point, and umbilical level) using a measuring tape in centimeters.
Duration of chest tube | Up to 1 week
  Duration of chest tube
Length of ICU stay | For up to 1 week
  Measure the duration of the patient's ICU stay
Hemodynamic Parameters | For the first three postoperative days
  Hemodynamic parameters will include oxygen saturation, which will be assessed using the pulse oximeter and will be expressed as a percentage %

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiothoracic and Vascular Surgery Center, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided